CLINICAL TRIAL: NCT01152047
Title: The Effect of Oxytocin on Satiety in Patients With Dyspepsia
Brief Title: The Effect of Oxytocin on Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Bodil Ohlsson, Department of Clinical Sciences, Division of Internal Medicine, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/502; 2009/502 (Other: Regional Ethical Review Board)
Record Dates: First submitted 2010-06-23; First posted 2010-06-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Dyspepsia; Lack of Satiety
Keywords: oxytocin; satiety; dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxytocin, satiety (Experimental): Oxytocin is given as infusion to examine if this decreases satiety compared to saline during a drinking test
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — 40mU/min as infusion of oxytocin
  Other Names: syntocinon

SUMMARY:
The investigators have seen that oxytocin lowers satiety in healthy subjects. Patients with dyspepsia suffers from decreased accommodation and increased satiety postprandially. The investigators now want to examine whether oxytocin may diminish symptoms in these patients.

DETAILED DESCRIPTION:
Patients will come twice for a slow satiety drinking test. Once they will get saline infusion and once oxytocin 40 mU/min. At the same time they register satiety on a VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* Dyspepsia

Exclusion Criteria:

* Age > 65 years
* Cardiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Satiety | 2 h
  The investigator want to examine whether oxytocin leads to lower satiety scores after intake of the same volume of nutrient

OTHER OUTCOMES:
To see if oxytocin lowers satiety | 2h
  To perform a drinking satiety test twice. Once with oxytocin and once with saline. Then examine whether oxytocin decreases satiety compared to saline

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Ohlsson, professor, Principal Investigator — Divsion of Internal Medicine
Locations (1):
- Skåne University Hospital, Malmo, Sweden